CLINICAL TRIAL: NCT02285712
Title: Contribution of Ultrasound for Peripheral Intravenous Catheter Placement by Intensive Care Nurses
Brief Title: Ultrasound-Guided Peripheral Intravenous Access by Critical Nurses.
Acronym: IDECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01143-44
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Venous Catheterization
Keywords: Peripheral venous catheter; ultrasound; nurse; Intensive Care Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Classical method of peripheral venous catheterization (No Intervention): Classical method will be applied only on arm and forearm.
- Ultrasound guided peripheral venous catheterization (Experimental): Nurse will use a vascular ultrasound system to orient the catheter toward the peripheral vein. Ultrasound method will be applied only on arm and forearm.
  Interventions: Device: Vascular ultrasound system

INTERVENTIONS:
Device: Vascular ultrasound system
  Arms: Ultrasound guided peripheral venous catheterization

SUMMARY:
Peripheral intravenous access is a major intervention in patients admitted to an intensive care unit. Systematically performed by nurses, it is also an essential intervention when the central venous access has to be removed. However, in the intensive care unit, patient centered-characteristics such as previous history of intravenous drug abuse, obesity, history of multiple vascular punctures or fluid overload most often affect the success rate of this procedure. For these patients, failure consequences are numerous: 1) delayed discharge from the intensive care unit, 2) increased pain and dissatisfaction, 3) increased incidence of catheter-related bloodstream infections. The use of ultrasound has gained increasing popularity particularly for obtaining central venous access. We hypothesize that, among trained nurses, ultrasound-guided peripheral venous access could represent an attractive alternative compared to the traditional anatomical method in order to increase the success rate.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted in ICU
* patient not able to express his opposition
* central venous access that need to be removed
* need for a peripheral venous access
* no clinical instability
* no visible superficial vein due to: BMI> 30, fluid overload, previous history of IV drug abuse, previous history of chemotherapy ,

Exclusion Criteria:

* patient < 18 yo
* pregnancy
* patient under protective supervision
* need for a central venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
number of peripheral venous catheterization attempts | up to day 2
  Each day, only 3 attempts are allowed

SECONDARY OUTCOMES:
Number of central lines removed | intraoperative
central venous catheter dwell time | intraoperative
  defined period between insertion and removal of the central venous line
peripheral venous catheter dwell time | intraoperative
  defined period between insertion and removal of the peripheral catheter with a maximum of 3 days.
number of central line catheter related infection | intraoperative
number of central line catheter related colonization | intraoperative
Diameter of the inserted peripheral venous catheter | day 0, or day 1 or day 2
  at peripheral venous catheter insertion
patient satisfaction | intraoperative
  assessed by an analogic scale
nurse satisfaction | intraoperative
  assessed by a survey form
Proportion of peripheral venous catheter successful placement | at day 0, day 1, day 2

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Kimmoun, M.D, Principal Investigator — Intensive care unit
Locations (1):
- CHU Nancy - Service de Réanimation Médicale Brabois, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Bridey C, Thilly N, Lefevre T, Maire-Richard A, Morel M, Levy B, Girerd N, Kimmoun A. Ultrasound-guided versus landmark approach for peripheral intravenous access by critical care nurses: a randomised controlled study. BMJ Open. 2018 Jun 9;8(6):e020220. doi: 10.1136/bmjopen-2017-020220. PMID 29886442